CLINICAL TRIAL: NCT01762059
Title: The Beacon Hill Study: Feasibility of Outpatient Automated Blood Glucose Control With a Bi-hormonal Bionic Endocrine Pancreas
Brief Title: Outpatient Automated Blood Glucose Control With a Bi-hormonal Bionic Endocrine Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012P002317
Record Dates: First submitted 2012-12-21; First posted 2013-01-07 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; continuous glucose monitoring; CGM; outpatient; insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bi-homonal Bionic Pancreas (Experimental): Closed-loop blood glucose control with a bi-hormonal bionic endocrine pancreas designed by Edward Damiano and Firas El-Khatib of Boston University. The device will deliver insulin lispro (Humalog) and glucagon based on blood glucose levels estimated by a continuous glucose monitoring device (Dexcom G4 Platinum) and a proprietary dosing algorithm. Blood glucose control will be automated for 5 days during which volunteers will sleep in a hotel and roam freely in downtown Boston during the day. There will be no restrictions on diet or exercise.
  Interventions: Device: Bi-homonal Bionic Pancreas
- Usual Care (Active Comparator): Usual care for 5 days (insulin pump therapy according to usual practice), volunteers will sleep at home and maintain their usual schedule during the day, there will be no restrictions on diet or exercise, they will wear a blinded CGM
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Bi-homonal Bionic Pancreas — A computer algorithm will automatically deliver insulin lispro and glucagon based on the signal from a minimally invasive continuous glucose monitor.
  Other Names: Boston University Bionic Pancreas
  Arms: Bi-homonal Bionic Pancreas
Other: Usual care
  Arms: Usual Care

SUMMARY:
This study will test the hypothesis that a wearable automated bionic pancreas system that automatically delivers both insulin and glucagon can improved glycemic control vs. usual in the outpatient environment.

DETAILED DESCRIPTION:
The study population will be volunteers with type 1 diabetes who are 21 years of age or older. The setting will be an outpatient environment in a three square-mile area on the Boston Peninsula (see Appendix A). Volunteers will stay in a hotel adjacent to the MGH campus at night and will have free activity during the day within the specified geographic area. They will determine the timing and nature of their meals from local restaurants, with food brought from home, or food kept in their hotel room, which will have a small refrigerator. They will have the opportunity to exercise as they wish in their choice of two gyms. There will be minimal scheduling constraints, limited only by an 11:00 PM curfew and morning departure time from the hotel of no earlier than 7:00 AM. They will be able to work if they wish as long as that can be done within the geographical constraints (e.g. if they work in the downtown Boston area or can "work from home" or have meetings at a conference room in the hotel or at a restaurant). During the entire experiment they will be closely monitored by study staff (RN, NP, or MD) around the clock. They will remain within direct line of sight and no more than a short distance away from study staff during the daytime for safety. During the night they will be continuously monitored via BG telemetry from a nearby hotel room and study staff will be able to enter their rooms quickly, should that become necessary. During the night, when volunteers will remain in their rooms, one study staff member will monitor up to two volunteers at a time.

Capillary BG will be tested every two hours during the day using a highly accurate, laboratory equivalent meter (HemoCue, selected for maximum data integrity) and venous BG will be tested every 30 minutes overnight using an autosampling device (GlucoScout). Continuous glucose monitoring (Dexcom G4) will be done throughout the study period. Photos and menu information, if available, will be documented for each meal and snack by the escort and estimates of carbohydrate intake will be estimated later from this information by a nutritionist. The type and level of activity being performed by the volunteers (e.g. lying, sitting, standing, walking, running) will be documented in 15 minute intervals by the study staff escort. Additional data will be collected using an accelerometer. During exercise, the type and duration of exercise, and, depending on the kind of activity, the heart rate (recorded using a Polar heart rate monitor) will be documented every 15 minutes and point-of-care blood glucose will be documented every 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older with type 1 diabetes for at least one year
* Stimulated C-peptide < 0.1 nmol/L at 90 minutes after liquid mixed meal by the DCCT protocol
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins including insulin aspart (NovoLog), insulin lispro (Humalog), and insulin glulisine (Apidra) for at least three months prior to enrollment
* Otherwise healthy (mild chronic disease such as asthma, hypertension, and depression will be allowed if well controlled)

Exclusion Criteria:

* Unable to provide informed consent
* Unable to comply with study procedures
* Total daily dose (TDD) of insulin that is > 1.5 U/kg
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception.
* Hypoglycemia unawareness (self-reported lack of hypoglycemia symptoms when BG is < 50 mg/dl)
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
* Any known history of coronary artery disease (CAD)
* Abnormal EKG suggestive of coronary artery disease or increased risk of malignant arrhythmia
* Congestive heart failure (established history of CHF, paroxysmal nocturnal dyspnea, or orthopnea).
* History of TIA or stroke.
* History of pheochromocytoma. Fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor
* Untreated or inadequately treated mental illness
* Current alcohol abuse or substance abuse
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference.
* Use non-insulin, injectable anti-diabetic medications or oral anti-diabetic medications
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Unwilling or unable to completely avoid acetaminophen
* ALT > 3-fold upper limit of normal
* Albumin < 3 g/dl
* Body mass index less than18 or greater than 35

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Russell SJ, El-Khatib FH, Sinha M, Magyar KL, McKeon K, Goergen LG, Balliro C, Hillard MA, Nathan DM, Damiano ER. Outpatient glycemic control with a bionic pancreas in type 1 diabetes. N Engl J Med. 2014 Jul 24;371(4):313-325. doi: 10.1056/NEJMoa1314474. Epub 2014 Jun 15. PMID 24931572
- See also: Information about this and related studies — http://www.artificialpancreas.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Bi-hormonal Bionic Pancreas and Usual Care: Closed-loop blood glucose control with a bi-hormonal bionic endocrine pancreas designed by Edward Damiano and Firas El-Khatib of Boston University. The device will deliver insulin lispro (Humalog) and glucagon based on blood glucose levels estimated by a continuous glucose monitoring device (Dexcom G4 Platinum) and a proprietary dosing algorithm. Blood glucose control will be automated for 5 days during which volunteers will sleep in a hotel and roam freely in downtown Boston during the day. There will be no restrictions on diet or exercise.
  After the first experimental period, there was a two-day washout period followed by the second experimental period.
  Usual care for 5 days (insulin pump therapy according to usual practice), volunteers will sleep at home and maintain their usual schedule during the day, there will be no restrictions on diet or exercise, they will wear a blinded CGM
  Usual care
Period: Overall Study
Arm/Group | All Participants: Bi-hormonal Bionic Pancreas and Usual Care
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Average Blood Glucose (Co-primary Outcome)
Description: Average blood glucose during the closed-loop control period as determined from HemoCue capillary measurements (daytime+nightime) and GlucoScout venous measurements (nighttime).
Time Frame: 5 days of closed-loop control
Population: This outcome measure was only assessed for the closed loop control period, and was not assessed during the usual care arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Bionic Pancreas: Closed loop blood glucose control using a bihormonal bionic endocrine pancreas delivering insulin and glucagon using continuous glucose monitor readings, with doses calculated by a computer algorithm every 5 minutes .
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 20
mg/dL | 138 (14)

2. Primary Outcome: Percentage of Time Blood Glucose Values Less Than 70 mg/dl (Co-primary Outcome)
Description: Percentage of time blood glucose values during the closed-loop control period less than 70 mg/dl determined from HemoCue capillary measurements (daytime) and GlucoScout venous measurements (nighttime) during day 1-5.
  During usual care (open loop), blood sugars were not checked through GlucoScout or HemoCue (as per usual care fashion) and so were not compared to bionic pancreas (closed loop) arm
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 20
percentage of time | 4.8 (5.2)

3. Secondary Outcome: Average BG During the Closed-loop Control Period as Determined From All HemoCue Measurements Taken During the Daytime and All Scheduled GlucoScout Measurements During the Nighttime.
Description: During usual care (open loop), blood sugars were not checked through GlucoScout or HemoCue (as per usual care fashion) and so were not compared to bionic pancreas (closed loop) arm
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bi-homonal Bionic Pancreas
Number analyzed (Participants) | 20
mg/dl | 138 (14)

4. Secondary Outcome: Percentage of the Subset of BG Values Less Than 70 mg/dl as Determined From All All HemoCue Measurements Taken During the Daytime and Scheduled GlucoScout Measurements Taken During the Nighttime.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | All Participants: Bi-hormonal Bionic Pancreas and Usual Care
Number analyzed (Participants) | 20
percentage of time | 4.8 (5.2)

5. Secondary Outcome: Difference in the Average BG Between the Closed-loop Control Period and the Usual Care Period.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Difference in the Percentage of the Above Subset of BG Values Between the Closed-loop Control and Usual Care Periods Less Than 70 mg/dl.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Subjects With Mean BG < 154 mg/dl.
Description: This outcome measure was only assessed for the closed loop control period, and was not assessed during the usual care arm.
Time Frame: 5 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 20
percentage of participants | 100

8. Secondary Outcome: Difference in the Percentage of Subjects With Mean BG < 154 mg/dl During the Closed-loop Period vs. the Usual Care Period.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Hypoglycemic Events as Determined From GlucoScout and HemoCue Measurements.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Nadir BG During Exercise.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Correlation Between Exercise Intensity and Likelihood of a Hypoglycemic Event
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Average BG During the Closed-loop Control Period as Determined From All GlucoScout Measurements Taken During the Nighttime Monitoring.
Description: as for outcome 7
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 20
mg/dl | 125 (19)

13. Secondary Outcome: Fraction of Time Spent Within Each of the Following Glucose Ranges as Determined From All GlucoScout and HemoCue Measurements.
Description: Measurements adjusted for the frequency of measurement (i.e. modeled so that more frequent measurements at the time of hypoglycemia and exercise will not skew the mean):
  < 70 mg/dl,70-120 mg/dl,70-180 mg/dl, >180 mg/dl, >250 mg/dl
Time Frame: 5 Days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Difference of Outcome Measures on Days 1-2 vs. on Remaining Days (Days 3-5) During the Closed-loop Period.
Time Frame: 5 Days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Mean BG During Exercise.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Hypoglycemic Episodes During Exercise.
Time Frame: 5 days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

17. Secondary Outcome: Difference of Outcome Measures on Day 1 vs. Remaining Days (Days 2-5) During the Closed-loop Period.
Time Frame: 5 Days
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

18. Other Pre Specified Outcome: Percentage of Subjects With Mean CGMG < 154mg/dl
Time Frame: 5 days
Measure: Number; unit: percentage of subjects
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 20 | 20
percentage of subjects | 100 | 45

19. Other Pre Specified Outcome: Difference in the Percentage of Subjects With Mean CGMG <154mg/dl During the Closed-loop Period vs. the Usual Care Period
Time Frame: 5 days
Measure: Number; unit: percentage of subjects
Arm/Group | All Participants
Number analyzed (Participants) | 20
percentage of subjects | 55

20. Other Pre Specified Outcome: Fraction of Time Spent Within Each of the Following Glucose Ranges: < 70 mg/dl,70-120 mg/dl,70-180 mg/dl,>180 mg/dl,>250 mg/dl
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 20 | 20
percentage of time
  <70mg/dL | 4.1 (3.5) | 7.3 (4.7)
  70-120mg/dL | 47.7 (10.5) | 30.8 (15.7)
  70-180mg/dL | 79.5 (8.3) | 58.8 (14.6)
  >180mg/dL | 16.5 (7.9) | 33.8 (16.4)

21. Other Pre Specified Outcome: Mean Blood Sugar as Measured by Continuous Glucose Monitor (CGM) Readings
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 20 | 20
mg/dL | 133 (13) | 159 (30.4)

ADVERSE EVENTS:
Time Frame: 12 days
Description: Adverse events were collected for the Bionic Pancreas period, and were not collected during the usual care period.
Arm/Group | Bionic Pancreas (Closed Loop)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bionic Pancreas (Closed Loop) (N=20)
Headaches (General disorders) | 3 — Headache occurred three times on two subjects on the bionic pancreas.
Nausea (Gastrointestinal disorders) | 4 — Nausea without vomiting occurred one time each in four subjects on the bionic pancreas. In three of these cases, no glucagon dosing had occurred in over 2 hours.
Vomiting (Gastrointestinal disorders) | 1 — Nausea with vomiting occurred in one subject in the setting of an intravenous catheter removal, with the last glucagon dosed approximately 1 hour earlier.
Pain (Skin and subcutaneous tissue disorders) | 3 — Three insulin infusion sets and one glucagon infusion set were removed for pain or inflammation during the bionic pancreas arm.
Ketones (Endocrine disorders) | 1 — One subject developed moderate hyperketonemia (0.8 mmol/l) on the bionic pancreas in the setting of a leaking insulin infusion set. The hyperketonemia resolved afterthe infusion set was changed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes